CLINICAL TRIAL: NCT05946252
Title: Acute Effect of Motor Imagery in High-Risk Pregnants: A Randomized Controlled Pilot Study
Brief Title: Motor Imagery in High-Risk Pregnants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Seda Yakit Yesilyurt, Lecturer Dr, Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: İEU_SYY_1
Record Dates: First submitted 2023-06-14; First posted 2023-07-14 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy, High Risk

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery Group (Experimental): Risky pregnant women who have completed the 12th week of pregnancy, received inpatient treatment and have any of the following risk factors will be included in the study:
  * Pregnant women who are at risk for obstetric outcomes such as cervical insufficiency, multiple pregnancy and uncontrolled gestational diabetes, and physical activity restriction is recommended due to these conditions, and exercise is contraindicated,
  * Pregnant women with a maternal body mass index above 30, which causes them to be physically inactive
  Interventions: Other: Motor imagery; Other: Diaphragmatic breathing
- Control Group (Active Comparator): Risky pregnant women who have completed the 12th week of pregnancy, received inpatient treatment and have any of the following risk factors will be included in the study:
  * Pregnant women who are at risk for obstetric outcomes such as cervical insufficiency, multiple pregnancy and uncontrolled gestational diabetes, and physical activity restriction is recommended due to these conditions, and exercise is contraindicated,
  * Pregnant women with a maternal body mass index above 30, which causes them to be physically inactive
  Interventions: Other: Diaphragmatic breathing

INTERVENTIONS:
Other: Motor imagery — Motor imagery will be performed according to the PETTLEP (Physical,Environment,Task,Time,Learn,Emotion,Perspective) model for 15 minutes.
  1. To imagine walking activity in different environments (seaside, beach, walking path).
  2. The rest activity will be imagined by sitting on a bench.
  3. Upper extremity strengthening exercises with dumbbells, lower extremity strengthening exercises with elastic band and trunk-oriented bridging, posterior pelvic tilt and table top stabilization exercises will be visualized.
  4. The rest activity will be imagined by sitting on a bench.
  5. Imagination will end with homecoming and domestic activities.
  Arms: Motor Imagery Group
Other: Diaphragmatic breathing — Diaphragmatic breathing will be shown to pregnant women in the supine position, eyes closed, with one hand on the chest and the other hand on the abdomen. This practice will last for five minutes.

SUMMARY:
The aim of this study is to determine the acute effects of motor imagery exercises on fetal heart rate, uterine contractions, maternal heart rate, blood pressure, oxygen saturation and well-being in high-risk pregnant women.

DETAILED DESCRIPTION:
Bed rest is often recommended in high-risk pregnant women to prevent complications from reaching dangerous levels.

Pregnant women recommended bed rest can benefit from exercise in order to overcome this process more easily, to reduce the negative consequences of inactivity and to prevent possible risks.

However, there may be differences between the view of high-risk pregnant women and the view of healthy pregnant women. Motor imagery refers to a mental process in which an individual mentally imagines that movement without actually eliciting an active movement. Studies have shown that similar brain regions are activated during movement performance and movement imagery. It has been reported in the literature that progressive relaxation exercises performed under mental/motor imagery guidance in healthy pregnant women and pregnant women lead to an improvement in maternal anxiety, stress and fetal attachment scales and a decrease in maternal systolic/diastolic blood pressure. However, as far as the investigators know, there is no study that applies the exercise protocol that can be given to healthy pregnant women to high-risk pregnant women with motor imagery and examines acute responses on fetal and maternal parameters.

ELIGIBILITY:
Inclusion Criteria:

Risky pregnant women who have completed the 12th week of pregnancy, received inpatient treatment and have any of the following risk factors will be included in the study:

* Pregnant women who are at risk for obstetric outcomes such as cervical insufficiency, multiple pregnancy and uncontrolled gestational diabetes, and physical activity restriction is recommended due to these conditions, and exercise is contraindicated,
* Pregnant women with a maternal body mass index above 30, which causes them to be physically inactive

Exclusion Criteria:

* Pregnant women who are at risk for obstetric outcomes such as gestational diabetes mellitus and pregnancy-induced hypertension, but physical activity is recommended
* Pregnant women with severe cardiovascular, pulmonary and systemic disorders
* Pregnant women with psychological seizure disorders
* Pregnant women who do not have any mental problems that prevent cooperation and understanding
* Pregnant women with any medical condition that prevents the safe and effective implementation of interventions.
* Pregnant women in other high-risk groups (such as early membrane rupture, placenta previa, preeclampsia) that may have early intervention in terms of obstetric outcomes.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Maternal self well-being | at baseline
  Well-being will be assessed on a numbered classification scale-11. '0' indicates worse self well-being, '10' indicates excellent self well-being.

SECONDARY OUTCOMES:
Maternal self well-being | immediately after intervention
  Well-being will be assessed on a numbered classification scale-11. '0' indicates worse self well-being, '10' indicates excellent self well-being.
Maternal heart rate | at baseline
  Heart rate measurements will be made with an arm type digital sphygmomanometer.
Maternal heart rate | in the 7th minutes of the intervention
  Heart rate measurements will be made with an arm type digital sphygmomanometer.
Maternal heart rate | immediately after intervention
  Heart rate measurements will be made with an arm type digital sphygmomanometer.
Maternal blood pressure (systolic pressure) | at baseline
  Blood pressure measurements will be made with an arm type digital sphygmomanometer.
  Systolic blood pressure and diastolic blood pressure will be assessed.
Maternal blood pressure (systolic pressure) | in the 7th minutes of the intervention
  Blood pressure measurements will be made with an arm type digital sphygmomanometer.
  Systolic blood pressure and diastolic blood pressure will be assessed.
Maternal blood pressure (systolic pressure) | immediately after intervention
  Blood pressure measurements will be made with an arm type digital sphygmomanometer.
  Systolic blood pressure and diastolic blood pressure will be assessed.
Maternal blood pressure (diastolic pressure) | at baseline
  Blood pressure measurements will be made with an arm type digital sphygmomanometer.
  Systolic blood pressure and diastolic blood pressure will be assessed.
Maternal blood pressure (diastolic pressure) | in the 7th minutes of the intervention
  Blood pressure measurements will be made with an arm type digital sphygmomanometer.
  Systolic blood pressure and diastolic blood pressure will be assessed.
Maternal blood pressure (diastolic pressure) | immediately after intervention
  Blood pressure measurements will be made with an arm type digital sphygmomanometer.
  Systolic blood pressure and diastolic blood pressure will be assessed.
oxygen saturation | at baseline
  Finger type pulse oximeter will be attached and peripheral oxygen saturation will be monitored.
oxygen saturation | in the 7th minutes of the intervention
  Finger type pulse oximeter will be attached and peripheral oxygen saturation will be monitored.
oxygen saturation | immediately after intervention
  Finger type pulse oximeter will be attached and peripheral oxygen saturation will be monitored.
Fetal Heart Rate | at baseline
  Fetal heart rate will be monitored with a cardiotachometer (Philips Avalon Fetal Monitor).
Fetal Heart Rate | in the 7th minutes of the intervention
  Fetal heart rate will be monitored with a cardiotachometer (Philips Avalon Fetal Monitor).
Fetal Heart Rate | immediately after intervention
  Fetal heart rate will be monitored with a cardiotachometer (Philips Avalon Fetal Monitor).
Uterine contractions severity | at baseline
  Uterine contractions severity will be monitored with a cardiotachometer (Philips Avalon Fetal Monitor).
Uterine contractions severity | in the 7th minutes of the intervention
  Uterine contractions severity will be monitored with a cardiotachometer (Philips Avalon Fetal Monitor).
Uterine contractions severity | immediately after intervention
  Uterine contractions severity will be monitored with a cardiotachometer (Philips Avalon Fetal Monitor).

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yakıt Yeşilyurt, PT, PhD, Principal Investigator — Izmir University of Economics
Locations (1):
- Health Sciences University İzmir Tepecik Education and Research Hospital Gynecology and Obstetrics Clinic, Izmir, Turkey (Türkiye)